CLINICAL TRIAL: NCT04470180
Title: An RCT of Virtual Teach-to-Goal Versus Brief Instruction for Children With Asthma in Clinics
Brief Title: Virtual Teach to Goal vs. Brief Intervention Inhaler Study-outpatient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: American Thoracic Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 192091
Record Dates: First submitted 2020-04-16; First posted 2020-07-14 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Asthma in Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Teach-to-Goal (V-TTG) (Experimental): They will be randomized to receive education via a virtual learning module.
  Interventions: Behavioral: Virtual Teach to Goal
- standardized brief intervention (Active Comparator): Intervention that mimics usual care to deliver inhaler technique education.
  Interventions: Behavioral: Brief Instruction

INTERVENTIONS:
Behavioral: Virtual Teach to Goal — Participants will complete inhaler education on a tablet device.
  Arms: Virtual Teach-to-Goal (V-TTG)
Behavioral: Brief Instruction — Participants will be read out loud instruction on how to use their inhaler.
  Arms: standardized brief intervention

SUMMARY:
This study aims to evaluate the comparative effectiveness of a high-fidelity, low-resource, and feasible model versus a standardized brief intervention that mimics usual care to deliver tailored inhaler technique education to children with asthma via a randomized clinical trial. We have already conducted a trial of V-TTG among elementary school-aged children hospitalized in the inpatient setting and we now aim to test this tool in the outpatient clinic setting among a broader pediatric patient population.

DETAILED DESCRIPTION:
Asthma is the most common chronic childhood condition and has significant adverse consequences. One in 12 United States children has asthma, resulting in 13.4 million missed school days, 1 million emergency department visits, and 140,000 hospitalizations annually. Urban, minority, and underserved youth are disproportionally affected. On Chicago's South Side, one-in-five children have an asthma diagnosis; over half visit an urgent care or emergency department (55%), miss school (51.2%), or require parents to miss work annually due to asthma (56.1%).

Effective self-management is crucial to optimize asthma care and improve outcomes. A key barrier to self-management is the improper use of respiratory inhalers, which limits disease control. Better inhaler technique is associated with improved asthma outcomes for children. Assessment and education of inhaler technique are recommended at all healthcare encounters; however, it is limited in practice because it is resource-intensive (both personnel and time) and lacks fidelity. Thus, low-resource interventions that accurately teach inhaler skills are needed to impact pediatric asthma outcomes.

Teach-to-Goal (TTG) is a patient-centered strategy that uses tailored rounds of teaching and assessments to ensure mastery of inhaler technique. Studies show it is effective but resource-intensive. A "virtual TTG" (V-TTG) intervention represents an opportunity to deliver inhaler technique education with a high-fidelity, low-resource, and feasible strategy. The module utilizes innovative learning technology with video demonstrations and assessment questions to tailor education to each user; the cycles of assessment and education continues until satisfactory mastery is achieved. Our team developed a V-TTG intervention for adults with demonstrated efficacy. It remains unknown whether this interactive and adaptive module will be feasible and effective in the pediatric population due to varied developmental levels and parental involvement in care.

Virtual Teach-to-Goal (V-TTG) holds the potential to improve inhaler technique in children; however, because learning theory indicates children and adults learn differently, the same learning module cannot be utilized. We have already constructed V-TTG for children with feedback from children with asthma, parents, and healthcare professionals. The learning module is tailored for age by using developmentally and age-appropriate vocabulary, concepts, format, and pacing.

ELIGIBILITY:
Inclusion Criteria:

* Families will be included in the study if:

  1. The child is between the ages of 6-17 years old
  2. The child has a diagnosis of asthma, wheezing, or bronchospasm
  3. The child has been or is seen in general pediatrics, pediatric pulmonary, or pediatric allergy clinic at the University of Chicago Medical Center
  4. The child is taking medication for asthma, wheezing, or bronchospasm (either a controller medication or a quick-relief medication)
  5. The family has acess to wifi and/or data that supports virtual video-based platforms (if study is done virtually)

Exclusion Criteria:

* Families will be excluded from the study if:

  1. The child/parent decline or unable to provide consent/assent
  2. The child/parent does not speak/read English
  3. The child cannot use an inhaler by themselves without a mask
  4. The child previously participated in this study
  5. The family does not have access to wifi and/or data that supports virtual video-based platforms (if study done virtually)

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2021-11-05 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with effective inhaler use (>75% steps correct) post-intervention with V-TTG versus BI | 12 months
  Inhaler technique will be assessed based on a validated published checklist, which was developed and validated by Dr. Press15 and utilized in my preliminary research with children (see Preliminary Studies). For this primary outcome, we will account for the pre-intervention technique to account for any differences in baseline of the two groups

SECONDARY OUTCOMES:
Number of inhaler technique steps correct pre- and post-V-TTG education | At baseline
  Evaluation of inhaler technique before and after education using validated checklist
Number of inhaler technique steps correct at 1 month | 1-month after enrollment
  Evaluation of inhaler technique 1-month after education/baseline session
Score of Asthma Control Survey | 12-months
  Assessed using validated survey measure
Score of Asthma Impact | 12-months
  Assessed using validated survey measure
Score of Caregiver Quality of Life | 12-months
  Assessed using validated survey measure
Score of Child Asthma Management Self-Efficacy | 12-months
  Assessed using validated survey measure
Number of healthcare encounters self-reported and EHR-recorded since baseline | 12-months
  Healthcare utilization measured via program-specific questionnaire delivered to parent and child as well as manual review of medical records

CONTACTS AND LOCATIONS:
Overall Officials: Anna Volerman, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No